CLINICAL TRIAL: NCT00838201
Title: An Open Label, Single Arm, Extension Study to Evaluate the Long Term Safety of Denosumab (AMG 162) in the Treatment of Bone Loss in Subjects Undergoing Androgen-Deprivation Therapy for Non-Metastatic Prostate Cancer
Brief Title: Extension Study to Evaluate Long Term Safety of Denosumab in Subjects Undergoing ADT for Non-Metastatic Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080537
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2013-09-24 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Cancer; Carcinoma; Castrate-Resistant Prostate Cancer; Prostate Cancer; Tumors
Keywords: Androgen deprivation therapy for non-metastatic prostate cancer
MeSH Terms: conditions — Neoplasms; Carcinoma; Prostatic Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — 60 mg SC of Denosumab will be administered on study day 1, month 6, month 12, and month 18

SUMMARY:
The purpose of this study is to describe the safety and tolerability of up to 5 years (ie, 3 years under the 20040138 Amgen study and 2 years on this study) denosumab administration as measured by adverse events, immunogenicity, and safety laboratory parameters in subjects who previously received denosumab for non-metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be currently participating in the 20040138 Amgen study
* Subjects must sign the informed consent before any study specific procedures are performed.

Exclusion Criteria

* Subjects with any prior diagnosis of bone metastasis
* Known hypocalcemia
* Developed sensitivity to mammalian cell derived drug products during the 20040138 study
* Currently receiving any investigational product other than denosumab or having received any investigational product during the 20040138 study
* Any disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2012-05-03 (Actual); Study Completion 2012-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (65):
- United States (26):
  - Research Site, Huntsville, Alabama
  - Research Site, Anaheim, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, San Bernardino, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Middlebury, Connecticut
  - Research Site, New Britain, Connecticut
  - Research Site, Trinity, Florida
  - Research Site, Fort Wayne, Indiana
  - Research Site, Greenbelt, Maryland
  - Research Site, Sartell, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Albany, New York
  - Research Site, Bay Shore, New York
  - Research Site, Garden City, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Lancaster, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Salem, Virginia
  - Research Site, Burien, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
- Canada (23):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, Brantford, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North Bay, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Finland (2):
  - Research Site, Seinäjoki
  - Research Site, Tampere
- Hungary (4):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Nyíregyháza
- Mexico (3):
  - Research Site, Mexico City, Distrito F
  - Research Site, Toluca
  - Research Site, Veracruz
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Siedlce
  - Research Site, Warsaw
  - Research Site, Wroclaw

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrollment date: 18 February 2009; Last subject enrollment date: 11 May 2010
Pre-assignment Details: Only recruited those who were participating in the safety follow-up of 20040138 study at the time, were willing to receive Denosumab, and met the inclusion/exclusion criteria. The first portion of the arm label indicates subjects' treatment groups (Placebo or Denosumab) in the parent study 20040138
Groups:
- Placebo/Denosumab 60 mg SC Q6M: Placebo in the parent study (NCT00089674), and denosumab 60 mg SC Q6M in the current study
- Denosumab/Denosumab 60 mg SC Q6M: Denosumab 60 mg SC Q6M in the parent study (NCT00089674), and denosumab 60 mg SC Q6M in the current study
Period: Overall Study
Arm/Group | Placebo/Denosumab 60 mg SC Q6M | Denosumab/Denosumab 60 mg SC Q6M
Started | 186 | 198
Completed | 144 | 145
Not Completed | 42 | 53
Not completed — Investigator decision, or other reasons | 2 | 3
Not completed — Noncompliance | 0 | 1
Not completed — Administrative decision | 1 | 2
Not completed — Disease progression | 3 | 3
Not completed — Consent withdrawn | 16 | 19
Not completed — Lost to Follow-up | 4 | 3
Not completed — Adverse Event | 5 | 9
Not completed — Death | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Denosumab 60 mg SC Q6M | Denosumab/Denosumab 60 mg SC Q6M | Total
Number analyzed (Participants) | 186 | 198 | 384
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73 (7.1) | 74.1 (6.6) | 73.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 186 | 198 | 384
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 153 | 173 | 326
  Black or African American | 6 | 8 | 14
  Hispanic or Latino | 26 | 17 | 43
  Japanese | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Through Month 24
Time Frame: 24 months
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Placebo/Denosumab 60 mg SC Q6M | Denosumab/Denosumab 60 mg SC Q6M
Number analyzed (Participants) | 186 | 198
Participants | 174 | 184

ADVERSE EVENTS:
Time Frame: about 38 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  One subject who was randomized to the placebo arm of the parent study received at least one dose of denosumab in the parent study and therefore was summarized in denosumab/denosumab arm.
Groups:
- Placebo/ Denosumab 60 mg Q6M: Placebo in the parent study (NCT00089674), and denosumab 60 mg SC Q6M in the current study
- Denosumab/ Denosumab 60 mg Q6M: Denosumab 60 mg SC Q6M in the parent study (NCT00089674), and denosumab 60 mg SC Q6M in the current study
Arm/Group | Placebo/ Denosumab 60 mg Q6M | Denosumab/ Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 45/185 | 51/199
Other Adverse Events (participants affected / at risk) | 47/185 | 46/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/ Denosumab 60 mg Q6M (N=185) | Denosumab/ Denosumab 60 mg Q6M (N=199)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 5 | 0
Cardiac ventricular disorder (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Sick sinus syndrome (Cardiac disorders) | 1 | 1
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Glaucoma (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Implant site haematoma (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Oxygen saturation abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 2
Convulsion (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 3
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/ Denosumab 60 mg Q6M (N=185) | Denosumab/ Denosumab 60 mg Q6M (N=199)
Constipation (Gastrointestinal disorders) | 16 | 13
Nausea (Gastrointestinal disorders) | 8 | 11
Urinary tract infection (Infections and infestations) | 6 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.